CLINICAL TRIAL: NCT01932333
Title: A Double-Blind, Placebo-Controlled, Randomized, Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-40411813 in Male and Female Elderly Subjects
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-40411813 in Male and Female Elderly Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017164; 40411813EDI1006 (Other: Johnson & Johnson Pharmaceutical Research & Development); 2010-019404-22 (EudraCT Number)
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Healthy; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; JNJ-40411813; Positive allosteric modulator
MeSH Terms: interventions — 1-butyl-3-chloro-4-(4-phenyl-1-piperidinyl)-(1H)-pyridone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: JNJ-40411813 50 mg; Drug: Placebo
- Cohort 2 (Experimental)
  Interventions: Drug: JNJ-40411813 100 mg; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-40411813 50 mg — Cohort 1: Participants will receive 50 mg of JNJ-40411813 (2 capsules X 25 mg) once a day on Day 1 in Period 1 and twice a day on Days 1 to 9 and once a day on Day 10 in Period 2 orally (by mouth).
  Arms: Cohort 1
Drug: JNJ-40411813 100 mg — Cohort 2: Participants will receive 100 mg of JNJ-40411813 (1 capsule X 100 mg) once a day on Day 1 in Period 1 and twice a day on Days 1 to 9 and once a day on Day 10 in Period 2 orally (by mouth).
  Arms: Cohort 2
Drug: Placebo — Cohort 1: Participants will receive placebo once a day on Day 1 for Period 1 and twice a day on Days 1 to 9 and once a day on Day 10 for Period 2; Cohort 2: Participants will receive placebo once a day on Day 1 for Period 1 and twice a day on Days 1 to 9 and once a day on Day 10 for Period 2.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (what the body does to the study medication) and pharmacodynamics (the study of the action or effects the study medication has on the body) of single- and multiple, escalating oral doses of JNJ-40411813.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor participants knows the treatment that the participant receives), randomized (study medication is assigned by chance), placebo-controlled (an inactive substance is compared with a medication to test whether the medication has a real effect in a clinical study), single- and multiple ascending dose study. This study consists of 3 phases: screening phase, treatment phase, and follow-up phase. This study will be conducted in 2 cohorts (groups) (Cohort 1: JNJ-40411813 50 mg and Cohort 2: JNJ-40411813 100 mg) and each cohort consists of 2 periods (Period 1: single dose and Period 2: multiple doses). Approximately 36 participants will be enrolled in this study (18 participants will be enrolled in each cohort) to receive JNJ-40411813 or placebo in 2:1 ratio. If safety/tolerability and pharmacokinetic results profile is favorable for single dose of JNJ-40411813, multiple dose administration will follow. Safety will be evaluated by the assessment of adverse events, vital signs, schellong test (a test for circulatory function), 12-lead electrocardiogram, physical examination, neurological examination (to measure mental status, motor examination, reflexes, sensory, gait and cranial nerves), vertigo (giddiness) symptom, and clinical laboratory tests which will be monitored throughout the study. The total duration of study participation for a participant will be 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must be postmenopausal for at least 12 months
* Body mass index (BMI) between 18 and 33 kg/m2 (BMI is calculated as weight [kilogram] divided by square of height [meter])

Exclusion Criteria:

* Clinically significant abnormal values for laboratory tests and abnormal physical examination
* Significant history of or current significant unstable medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, bronchospastic respiratory disease, dyspnea (difficulty in breathing), diabetes mellitus, thyroid disease, infection
* Significant history of or current psychiatric or neurological illness
* Serology positive for hepatitis B surface antigen, hepatitis C antibodies or HIV antibodies at screening
* Positive urine screen for drugs of abuse and positive alcohol breath test at screening or administration of the study medication
* Only the use of any prescription medication that is known to be potent CYP3A4 inhibitors or inducers within 2 weeks of start of study medication

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Cohort 1 and Cohort 2: Number of participants with adverse events | 9 weeks
Peak plasma concentration of JNJ 40411813 | Both Cohorts, Period 1: Day 1 (predose to 12 hrs), Day 2 (24 and 36 hrs), Day 3, and Day 4; Both Cohorts, Period 2: Day 1 (predose to 12 hrs); predose on Days 2, 3, 4, 5, 6, 7, 8, 9; Day 10 (predose to 12 hrs); Day 11 (0 and 12 hrs); Days 12, 13, and 14
  This sample will be used for pharmacokinetics analysis.
Time to reach the peak plasma concentration of JNJ 40411813 | Both Cohorts, Period 1: Day 1 (predose to 12 hrs), Day 2 (24 and 36 hrs), Day 3, and Day 4; Both Cohorts, Period 2: Day 1 (predose to 12 hrs); predose on Days 2, 3, 4, 5, 6, 7, 8, 9; Day 10 (predose to 12 hrs); Day 11 (0 and 12 hrs); Days 12, 13, and 14
  This sample will be used for pharmacokinetics analysis.
Area under the plasma concentration of JNJ 40411813 - time curve from 0 to t hours post dosing | Both Cohorts, Period 1: Day 1 (predose to 12 hrs), Day 2 (24 and 36 hrs), Day 3, and Day 4; Both Cohorts, Period 2: Day 1 (predose to 12 hrs); predose on Days 2, 3, 4, 5, 6, 7, 8, 9; Day 10 (predose to 12 hrs); Day 11 (0 and 12 hrs); Days 12, 13, and 14
  Time 't' is the time of the last quantifiable concentration of JNJ-40411813. This sample will be used for pharmacokinetics analysis.
Elimination rate constant of JNJ 40411813 | Both Cohorts, Period 1: Day 1 (predose to 12 hrs), Day 2 (24 and 36 hrs), Day 3, and Day 4; Both Cohorts, Period 2: Day 1 (predose to 12 hrs); predose on Days 2, 3, 4, 5, 6, 7, 8, 9; Day 10 (predose to 12 hrs); Day 11 (0 and 12 hrs); Days 12, 13, and 14
  This sample will be used for pharmacokinetics analysis.
Terminal half-life of JNJ 40411813 | Both Cohorts, Period 1: Day 1 (predose to 12 hrs), Day 2 (24 and 36 hrs), Day 3, and Day 4; Both Cohorts, Period 2: Day 1 (predose to 12 hrs); predose on Days 2, 3, 4, 5, 6, 7, 8, 9; Day 10 (predose to 12 hrs); Day 11 (0 and 12 hrs); Days 12, 13, and 14
  This sample will be used for pharmacokinetics analysis.
Area under the plasma concentration of JNJ 40411813 - time curve from 0 to infinity post dosing | Both Cohorts, Period 1: Day 1 (predose to 12 hrs), Day 2 (24 and 36 hrs), Day 3, and Day 4
  This sample will be used for pharmacokinetics analysis.
Predose plasma concentration of JNJ 40411813 | Both Cohorts, Period 2: Day 1 (predose to 12 hrs); predose on Days 2, 3, 4, 5, 6, 7, 8, 9; Day 10 (predose to 12 hrs); Day 11 (0 and 12 hrs); Days 12, 13, and 14
  This sample will be used for pharmacokinetics analysis.
Average plasma concentration of JNJ 40411813 at steady state | Both Cohorts, Period 2: Day 1 (predose to 12 hrs); predose on Days 2, 3, 4, 5, 6, 7, 8, 9; Day 10 (predose to 12 hrs); Day 11 (0 and 12 hrs); Days 12, 13, and 14
  This sample will be used for pharmacokinetics analysis.
Cognitive test | Both Cohorts, Period 1: Screening; Both Cohorts, Period 2: Day -1 (1 day before study treatment) and Day 7
  This test will be used for pharmacodynamics analysis. Cognitive test is a group of mental processes that includes attention, memory, producing and understanding language, learning, reasoning, problem solving, and decision making. It is assess by word presentation, immediate word recall, picture presentation, simple reaction time, digit vigilance, choice reaction time, spatial working memory, numeric working memory, delayed word recall, word recognition, and picture recognition. It refers to an information processing view of a participant's psychological functions.
Addiction Research Center Inventory questionnaire (ARCI-Q) | Both Cohorts, Period 1: Day -1 and Day 1 (3 hrs post dose); Both Cohorts, Period 2: Day 7
  This questionnaire will be used for pharmacodynamics analysis. The ARCI-Q is a 49-item questionnaire that probes subjective feeling induced by a drug and categorizes them in four classes of drugs of abuse (morphine-like opioids, alcohol, stimulants and hallucinogens). This test is a self-rating scale. Only 'True (positive)' responses are scored. One point is given for each true response in items. The final score is the sum of the total 'true' responses. Lower scores indicate worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Antwerp, Belgium